CLINICAL TRIAL: NCT04303221
Title: Effects of the Anchor System in the Postural Stability of Women Submitted to the Treatment of Breast Cancer
Brief Title: Effects of the Anchor System in the Postural Stability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Elaine Caldeira de Oliveira Guirro (Other)
Responsible Party: Sponsor-Investigator, Elaine Caldeira de Oliveira Guirro, Clinical professor, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3474028/2019
Record Dates: First submitted 2020-03-03; First posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer; Balance; Distorted
Keywords: Breast cancer; Lymphedema; Postural balance; Falls
MeSH Terms: conditions — Breast Neoplasms; Lymphedema | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GAJL - Young adult with lymphedema (Experimental): Women age 35 to 59 years (young adult) with lymphedema - exercise group
  Interventions: Other: Exercise
- GAJ - Young adult without lymphedema (Experimental): Women age 35 to 59 years (young adult) without lymphedema - exercise group
  Interventions: Other: Exercise
- GIL - Elderly with lymphedema (Experimental): Women aged 60 to 80 years (elderly) with lymphedema - exercise group
  Interventions: Other: Exercise
- GI - Elderly without lymphedema (Experimental): Women aged 60 to 80 years (elderly) without lymphedema - exercise group
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — The exercises will be performed three times a week (Mondays, Wednesdays and Fridays), lasting 60 min, 10 minutes of warm-up, 40 min of multisensory exercises, and 10 min of final relaxation, for 12 weeks.

SUMMARY:
Evaluate the effect of a balance rehabilitation program associated or not with the use of the anchor system, on the postural control of women undergoing breast cancer treatment.

DETAILED DESCRIPTION:
The aim of this study is to compare the effects of an exercise program associated or not with a non-rigid instrument, called the anchor system, on the postural control of women undergoing breast cancer treatment. For this purpose, 80 women submitted to breast cancer treatment will be invited to participate, divided into four homogeneous groups, determined by the sample calculation: women submitted to breast cancer treatment in the age group of 35 to 59 years (young adult) with lymphedema (GAJL), women in the same age group without lymphedema (GAJ), women in the age group 60 to 80 years (elderly) with lymphedema (GIL), and women in the same age group without lymphedema (GI). Cognitive status will be assessed by the Mini Mental State Examination. To assess the subsystems responsible for maintaining balance, the Balance Evaluation Systems Test (BESTest) will be used, presented in order to guide clinical intervention, in addition to the Falls Efficacy Scale -International (FES-I). The distribution of plantar pressure and balance will be assessed using baropodometry. For data analysis, a normality test and data distribution will be performed, in addition to a statistical test consistent with the appropriate intra and intergroup comparisons, with a significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing treatment for breast cancer, in the 35 to 59 age group with lymphedema, women in the same age group without lymphedema, women in the 60 to 80 age group with lymphedema, and women in the same age group without lymphedema.

Exclusion Criteria:

* Women diagnosed with rheumatic-orthopedic diseases; with complaints of balance; with injury to the peripheral nervous system of upper or lower limbs.

Ages: 35 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Functional balance | 5 minutes
  Balance evaluation systems test - BESTest
Accidental falls | 5 minutes
  Falls efficacy scale international - FES-I
Plantar pressure distribution | 10 minuntes
  Baropodometry system

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Guirro, PhD, Principal Investigator — University of Sao Paulo - Ribeirao Preto - Brazil
Locations (1):
- Medical School of Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rangon FB, Marinho IL, Cuviena CF, de Moraes R, de Jesus Guirro RR, de Oliveira Guirro EC. Effects of the Anchor System on Postural Balance of Women Undergoing Breast Cancer Treatment: A Clinical, Randomized, Controlled, and Crossover Trial. Arch Phys Med Rehabil. 2024 Feb;105(2):258-267. doi: 10.1016/j.apmr.2023.07.005. Epub 2023 Jul 25. PMID 37499853